CLINICAL TRIAL: NCT06226506
Title: Comparative Pharmacokinetic Study of Aprepitant Injection in Humans
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Cao Yu, Director of Clinical Trials Center of Affiliated Hospital of Qingdao University, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QLG2174-101
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Healthy
MeSH Terms: interventions — Aprepitant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (T)-Reference (R) (Experimental): In this trial, 24 healthy subjects are planned to be enrolled in fasting. According to the randomization table, subjects will be randomly assigned to the Group A: Test (T)-Reference (R), The washout period (dosing interval) between doses will be at least 7 days. After fasting for at least 10 hours.
  Interventions: Drug: Test (T) Aprepitant injection; Drug: Reference (R) Aprepitant injection
- Reference (R)-Test (T) (Experimental): In this trial, 24 healthy subjects are planned to be enrolled in fasting. According to the randomization table, subjects will be randomly assigned to the Group B: Reference (R)-Test (T), The washout period (dosing interval) between doses will be at least 7 days. After fasting for at least 10 hours.
  Interventions: Drug: Test (T) Aprepitant injection; Drug: Reference (R) Aprepitant injection

INTERVENTIONS:
Drug: Test (T) Aprepitant injection — Specification: Aprepitant injection 4.4ml∶32mg. Produced and supplied by Qilu Pharmaceutical (Hainan) Co.
Drug: Reference (R) Aprepitant injection — Specification: Aprepitant injection 4.4ml∶32mg. Produced by Heron Therapeutics, Inc and supplied by Qilu Pharmaceutical (Hainan) Co.

SUMMARY:
This is a single-center, open, randomized, single-dose, two-cycle, two-sequence, crossover pharmacokinetic study in healthy adult subjects.

The trial is planned to enroll 24 healthy subjects. Subjects will be randomized to one of two groups (Group A: T-R, Group B: R-T) according to the randomization table. The washout period (dosing interval) between doses will be at least 7 days. For example, for a washout period of 7 days, all subjects will receive the appropriate drug according to the randomized schedule on Day 1 of Cycle 1 and Day 8 of Cycle 2 of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an informed consent form before the trial and fully understand the content, process and possible adverse effects of the trial； 2. Ability to complete research in accordance with the requirements of the pilot program； 3. Subjects (including male subjects) who have been using effective contraception for 14 days prior to the first dose and who are willing to voluntarily use effective contraception from the time of signing the information until 6 months after the last dose without pregnancy, sperm or egg donation program； 4. Male and female subjects aged 18-45 years (both 18 and 45 years)； 5. Body mass index (BMI) within the range of 19.0~26.0kg/m2 (including threshold values) .

-

Exclusion Criteria:

1. Have a history of serious medical problems of the heart, liver, kidneys, gastrointestinal tract, nervous system, endocrine system, respiratory system, or mental abnormality, which in the opinion of the researcher are not suitable for the participant；
2. Abnormalities of clinical significance as determined by the clinician, including physical examination, vital signs, electrocardiogram, or clinical laboratory testing；
3. People with a history of specific allergies (asthma, etc.) or current allergic diseases (hives, eczema, etc.), or allergies (e.g., allergies to two or more medications, foods such as milk, or pollen), or allergies to any of soy, alcohol, or eggs, or known allergies to the components of this medication or to similar substances；
4. Women who are pregnant or breastfeeding, or who have a positive pregnancy test, or who are using long-acting contraceptives or contraceptive implants；
5. Positive for any one or more of the following: Hepatitis B Surface Antigen, Hepatitis C Antibody, HIV Antibody, or Syphilis Antibody；
6. History of substance abuse within five years, or drug use within 3 months prior to screening, or a positive urine drug screen；
7. Persons who have consumed an average of more than 14 units of alcohol (1 unit = 360milliliter of beer or 45milliliter of 40% alcohol by volume spirits or 150milliliter of wine) per week in the 3 months prior to screening, or who have been unable to stop alcohol intake from 24h prior to dosing until completion of blood sampling in that cycle, or who have had a positive breathalyzer test for alcohol；
8. Those who smoked an average of more than 5 cigarettes per day in the 3 months prior to screening or who refused to stop using tobacco products during the stay；
9. History of surgical procedure within 3 months prior to screening, or planned surgery during the study period；
10. Blood donation or massive blood loss (>400milliliter, except physiologic blood loss in women) within 3 months prior to administration, or platelet donation of ≥2 therapeutic doses within 1 month；
11. Participation in a clinical trial of any drug that was administered within the 3 months prior to administration；
12. Those who have used any prescription medication within 14 days prior to dosing；
13. Those who have used any over-the-counter medications, herbs, or supplements within 7 days prior to dosing；
14. Pimozide or any other drug that inhibits or induces hepatic metabolism (e.g., inducers - barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; depressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative-hypnotics, verapamil, fluoroquinolones, antihistamine) used within the last 30 days prior to administration. (including verapamil, fluoroquinolones, antihistamines)；
15. Those who have taken special diets (e.g., grapefruit and grapefruit-containing products), or had strenuous exercise, or other factors affecting the absorption, distribution, metabolism, or excretion of the drug within 48 hours prior to the administration of the drug；
16. Anyone who has consumed any xanthine-rich food (e.g. coffee, tea, chocolate, cocoa, milk tea, etc.) in the 48h prior to administration；
17. Those who have difficulty collecting blood, or who cannot tolerate venipuncture, or who have a history of blood or needle-sickness；
18. Subjects judged by other investigators to be unsuitable for participation. -

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-23 (Estimated); Primary Completion 2024-01-25 (Estimated); Study Completion 2025-01-25 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 72 hours
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC0-t) | 72 hours
  Area under the drug concentration-time curve from time 0 to the last accurately measurable concentration at sample collection time t
Area under the plasma concentration versus time curve (AUC0-∞) | 72 hours
  Area Under the Plasma Drug Concentration-Time Curve from Time 0 to Infinite Time